CLINICAL TRIAL: NCT00267683
Title: A Clinical Trial to Study the Efficacy and Safety of Insulin Aspart Three Times Per Day Compared to Glibenclamide Once or Twice Daily in Type 2 Diabetes by Comparison of Ability to Control Blood Glucose
Brief Title: Efficacy and Safety of Insulin Aspart Versus Glibenclamide in Type 2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This trial was terminated due to low recruitment
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANA-1667; JapicCTI-060200 (Registry Identifier: JAPIC)
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin aspart
Drug: glibenclamide

SUMMARY:
This trial is conducted in Japan. This is a clinical trial to study the efficacy and safety of thrice daily Insulin Aspart compared to Glibenclamide in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Diet therapy for at least 12 weeks, or diet therapy and oral hypoglycaemic agent(s) other than SU agents for at least 12 weeks
* No previous treatment with insulin and/or SU agents
* HbA1c between 7.5% and 10.0%
* Body Mass Index (BMI) below 30.0 kg/m2

Exclusion Criteria:

* Proliferative retinopathy or maculopathy requiring acute treatment
* Impaired hepatic function
* Impaired renal function
* Cardiac diseases
* Uncontrolled hypertension
* Known hypoglycaemia unawareness or recurrent major hypoglycaemia
* Current treatment with systemic corticosteroids

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-12; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 24 weeks of treatment

SECONDARY OUTCOMES:
Plasma glucose levels
Percentage of subjects achieving the treatment target of HbA1c value < 6.5%

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com